CLINICAL TRIAL: NCT04675346
Title: Exploring Unmet Needs and Attitudes to Skin Self-examination in Melanoma Survivors
Acronym: EUNASS
Status: Completed | Type: Observational
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Barts & The London NHS Trust (Other); Ninewells Hospital (Other); University of Oxford (Other)
Responsible Party: Principal Investigator, Rubeta Matin, Primary Investigator, Oxford University Hospitals NHS Trust
Other Study IDs: 19/SC/0554; 261224 (Other: IRAS)
Record Dates: First submitted 2020-12-15; First posted 2020-12-19 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Melanoma, Stage I; Melanoma Stage III; Melanoma, Stage II
MeSH Terms: conditions — Melanoma | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Questionnaire: The EUNASS Study Questionnaire is an electronic questionnaire (using the Qualtrics programme) designed to assess management after diagnosis of melanoma and during follow-up, health status, fear of melanoma recurrence, melanoma-specific supportive care needs, sun protection behaviour, views and habits about SSE and standard socio-demographic details.
  Interventions: Other: Questionnaire
- Interviews: A qualitative researcher will undertake 25-30 semi-structured interviews with participants who have volunteered their contact details in the final section of the EUNASS Study Questionnaire. A purposive sampling approach will be taken for participant recruitment to this part of the study.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire

SUMMARY:
This is a prospective, multi-centred cohort study whereby the EUNASS Study questionnaire will be administered electronically to identify needs of melanoma survivors, the extent to which these needs are being met, and identify areas which have the greatest need for development. It will also evaluate behaviour in relation to sun protection and skin self-examination (SSE). It will be a self-completed questionnaire.

Qualitative work using semi-structured interviews will explore the needs of melanoma survivors in greater depth, will present examples of potential interventions to improve SSE and explore factors that determine the likelihood of engaging in an intervention which can address unmet needs, such as improving SSE. Taken together, the data will provide the evidence base to inform the development of an intervention to improve SSE, which can subsequently be tested in secondary care services.

ELIGIBILITY:
Inclusion Criteria:

Participant is willing and able to give informed consent for participation in the study.

* Male or Female, aged 18 years or above.
* Histological diagnosis of primary cutaneous invasive melanoma (any Breslow thickness) at 3 - 12 months from diagnosis (as most primary treatment will be complete by 3 mths)
* American Joint Cancer Committee Version 8 [2018] (AJCC V8) Stage I - III melanoma at time of recruitment
* Able to complete an electronic questionnaire

Exclusion Criteria:

* Other current active internal malignancy (i.e. does not include non-melanoma skin cancers)
* Inability to independently complete electronic questionnaire
* AJCC V8 Stage IV melanoma at time of recruitment
* Clinical stage of disease unknown / unconfirmed

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending the Dermatology or Medical Oncology departments with a confirmed diagnosis of AJCC V8 stage I - III melanoma in the last year
Sampling Method: Non-Probability Sample
Enrollment: 252 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Mixed methods: analysis of a) Patient questionnaire responses and b) Semi-structured interviews | 2 years
  Mixed methods analysis - quantitative and qualitative results

CONTACTS AND LOCATIONS:
Overall Officials: Rubeta Matin, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Churchill Hospital, Headington, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No plan